CLINICAL TRIAL: NCT01825239
Title: Virtual Left Ventricular Lead Navigation in Patients With Ischemic Cardiomyopathy
Brief Title: Virtual LV Lead Navigation in Patients With Ischemic Cardiomyopathy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Problems with execution
Sponsor: University of Pittsburgh (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, David Schwartzman, Professor of Medicine, Cardiac Electrophysiology, University of Pittsburgh, University of Pittsburgh
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PRO12070339
Record Dates: First submitted 2013-04-02; First posted 2013-04-05 (Estimated); Last update posted 2015-08-07 (Estimated); Status verified 2015-08

CONDITIONS: Cardiomyopathy; Ischemic Cardiomyopathy
Keywords: ischemic cardiomyopathy; cardiomyopathy; left ventricular lead; cardiac electrophysiologic studies
MeSH Terms: conditions — Cardiomyopathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrophysiology Study (Other): This is a single arm study, all study participants will be referred for an Electrophysiology Study
  Interventions: Other: Collection of measurements during LV pacing during electrophysiology study

INTERVENTIONS:
Other: Collection of measurements during LV pacing during electrophysiology study — During the electrophysiology study, measurements will be obtained while pacing from different left ventricular regions in context to scar as determined by SPECT-CT testing.

SUMMARY:
Presently, the left ventricular lead is placed in a similar position for all patients. It is not known whether placing this lead in different positions in the heart will make the heart pump better. In this study, the investigator will collect measurements of the heart's electrical activity during an Electrophysiology Study (EP study or EPS). The hope is that these measurements will provide the know how to develop an individualized left ventricular lead placement "prescription" for patients referred for left ventricular lead pacing.

ELIGIBILITY:
Inclusion Criteria:

* Ischemic cardiomyopathy
* Intrinsic QRS duration >120 milliseconds
* LV ejection fraction <40%

Exclusion Criteria:

* Persistent atrial tachyarrhythmia
* Active cardiac ischemia
* Cerebrovascular accident within 6 months
* Surgical or percutaneous cardiac revascularization procedure within 3 months
* Under 18 years of age
* Pregnant
* Participating in a clinical study that would preclude enrollment
* Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-04; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
dP/dt measurements observed during pacing from different left ventricular regions | Measurements will be observed at the time of the electrophysiology study (EPS) at enrollment.
  During the electrophysiology study, the dP/dt measurements will be observed during pacing from different left ventricular regions.

CONTACTS AND LOCATIONS:
Overall Officials: David S. Schwartzman, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Hayes, D.L, et al. Resynchronization and Defibrillation for Heart Failure: A Practical Approach. UK: Blackwell Publishing, 2004.
- [Background] Ellenbogen K.A., et al. Device Therapy for Congestive Heart Failure. Pennsylvania: Saunders, 2004.
- [Background] Szydlo K, Wita K, Trusz-Gluza M, Urbanczyk D, Filipecki A, Orszulak W, Tabor Z, Krauze J, Kwasniewski W, Myszor J, Turski M, Kolasa J, Szczogiel J. Impact of left ventricular remodeling on ventricular repolarization and heart rate variability in patients after myocardial infarction treated with primary PCI: prospective 6 months follow-up. Ann Noninvasive Electrocardiol. 2008 Jan;13(1):8-13. doi: 10.1111/j.1542-474X.2007.00195.x. PMID 18234001
- [Background] Cohn JN, Ferrari R, Sharpe N. Cardiac remodeling--concepts and clinical implications: a consensus paper from an international forum on cardiac remodeling. Behalf of an International Forum on Cardiac Remodeling. J Am Coll Cardiol. 2000 Mar 1;35(3):569-82. doi: 10.1016/s0735-1097(99)00630-0. PMID 10716457
- [Background] S. Goel. Pacing For Patients With Congestive Heart Failure and Dilated Cardiomyopathy www.dcmsonline.org February, 2002/ Jacksonville Medicine
- [Background] Adelstein EC, Saba S. Scar burden by myocardial perfusion imaging predicts echocardiographic response to cardiac resynchronization therapy in ischemic cardiomyopathy. Am Heart J. 2007 Jan;153(1):105-12. doi: 10.1016/j.ahj.2006.10.015. PMID 17174647
- [Background] Barold SS, Herwerg B. Pacing in heart failure: how many leads and where? Heart. 2008 Jan;94(1):10-2. doi: 10.1136/hrt.2007.119404. No abstract available. PMID 18083947
- [Background] Schwartzman D, et al. Image-guided left ventricular pacing. Europace 2010; 12: 877-81.